CLINICAL TRIAL: NCT06463028
Title: An Open-label, Multi-Center, Phase 2 Clinical Trial Evaluating Sapanisertib and Serabelisib (PIKTOR) With Paclitaxel, and a Substudy Evaluating PIKTOR With Paclitaxel Plus an Insulin-Suppressing Diet, in Patients With Advanced or Recurrent Endometrial Cancer
Brief Title: Sapanisertib and Serabelisib (PIKTOR) With Paclitaxel and a Substudy With an Insulin-Suppressing Diet in Patients With Advanced/Recurrent Endometrial Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Faeth Therapeutics (Industry)
Collaborators: GOG Foundation (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FTH-PIK-201; GOG-3111 (Other: GOG Foundation/Partners)
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Endometrial Cancer
Keywords: Serabelisib; Sapanisertib; Paclitaxel; Taxol; Antineoplastic Agents; PI3K; AKT; mTOR; Dual PI3K/mTOR inhibition; Genetic mutation; Cisplatin; Carboplatin; Genital Diseases; Endometrial Neoplasms; Advanced Endometrial Carcinoma; Recurrent Endometrial Carcinoma; Metastatic Endometrial Carcinoma; Endometrial Cancer; Endometrioid Carcinoma; Cancer of Endometrium; Cancer of the Endometrium; Carcinoma of Endometrium; Endometrial Carcinoma; Endometrium Cancer; Neoplasms, Endometrial; Metabolism; Synthetic Lethality; Metabolism Programming; PIK3CA; PIK3CA Mutation; PI3K Gene Mutation; PI3K/AKT/mTOR Pathway Mutation; AKT Gene Mutation; mTOR Gene Mutation
MeSH Terms: conditions — Endometrial Neoplasms; Genital Diseases; Carcinoma, Endometrioid; Hereditary Sensory and Autonomic Neuropathies | interventions — sapanisertib; serabelisib; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- sapanisertib and serabelisib (PIKTOR) with paclitaxel (Experimental): Subjects will receive doses of sapanisertib and serabelisib (PIKTOR) administered orally and paclitaxel administered intravenously.
  Interventions: Drug: Sapanisertib; Drug: Serabelisib; Drug: Paclitaxel

INTERVENTIONS:
Drug: Sapanisertib — Oral
  Other Names: FTH-003; MLN0128
Drug: Serabelisib — Oral
  Other Names: FTH-001; MLN1117
Drug: Paclitaxel — Infusion

SUMMARY:
This is a Phase 2, multicenter, open-label, single-arm study to evaluate the efficacy and safety of sapanisertib and serabelisib (PIKTOR) with paclitaxel in participants with advanced or recurrent endometrial cancer.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, open-label, single-arm study to evaluate the efficacy and safety of sapanisertib and serabelisib (PIKTOR) with paclitaxel in participants with advanced or recurrent endometrial cancer who have failed prior systemic therapies, including a platinum-based therapy and an immune checkpoint inhibitor, either separately or together.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of endometrioid endometrial carcinoma.
* Documented evidence of advanced or recurrent endometrial cancer that is not amenable to surgery/radiation for curative intent.
* Participant has received at least 1 but not more than 4 prior systemic therapies. Prior therapy must include platinum-based chemotherapy and a checkpoint inhibitor, either separately or in combination. If a subject has been unable to be treated with checkpoint inhibitor in the past due to medical contraindications, consult with Medical Monitor.
* PI3K/AKT/mTOR pathway gene alteration identified.
* At least 1 measurable target lesion according to RECIST v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1 at Screening.
* Non-pregnant, non-lactating females who are postmenopausal, surgically sterile or who agree to use effective contraceptive methods..

Exclusion Criteria:

* Participants with central nervous system metastases are not eligible, unless they have completed local therapy and have discontinued the use of corticosteroids for this indication for at least 4 weeks before starting treatment in this study
* Active malignancy (except for endometrial cancer, definitively treated in-situ carcinomas [e.g., breast, cervix, bladder], or basal or squamous cell carcinoma of the skin) within the past 24 months prior to treatment. Fully resected localized malignancies are eligible.
* Gastric feeding tube (gastrostomy tube), gastrointestinal malabsorption, gastrointestinal anastomosis, bowel obstruction, or any other condition that might affect the absorption of study treatment.
* Clinically significant (per Investigator judgement) hemoptysis or tumor bleeding.
* Significant cardiovascular impairment.
* Active, uncontrolled (requiring systemic antimicrobial therapy) infection.
* Concurrent participation in another therapeutic clinical trial.
* Prior radiation therapy within 21 days prior to start of study treatment.
* Strong CYP3A4 inhibitors and inducers are prohibited during the study. Strong CYP1A2 inhibitors as well as CYP1A2 inducers should be administered with caution and at the discretion of the Investigator. Alternative treatments, if available, should be considered. Additionally, strong CYP3A4 inhibitors or inducers should not be taken within 7 days before the first dose of study intervention.
* Participants who require PPIs or chronic use of antacids, histamine H2 receptor blockers, or other treatments to raise gastric pH.
* Prolongation of QTc interval to >480 ms.
* HbA1c ≥ 8.0% or fasting serum glucose > 160 mg/dL or fasting triglycerides > 300 mg/dL or receiving treatment with insulin.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-12 (Actual); Primary Completion 2028-09 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | Up to 2 years
  Defined as the proportion of participants with measurable disease at baseline who have confirmed complete response (CR) or partial response (PR).

SECONDARY OUTCOMES:
Progression free survival (PFS) | Up to 5 years.
  Defined as the time from first dose until the date of disease progression or death.
Progression free survival (PFS) at 6 months | Up to 5 years.
  Defined as PFS rate at 6 months.
Overall survival (OS) | Up to 5 years.
  Defined as the time from first dose to death.
Clinical benefit rate (CBR) | Up to 5 years.
  Defined as the percentage of participants who achieve complete response (CR), partial response (PR), or have stable disease (SD) of at least 16 or 24 weeks.
Duration of response (DoR) | Up to 5 years.
  Defined for participants with confirmed CR or PR as the time from response until date of documented disease progression or death.
Safety and tolerability of drugs by assessment of adverse events (AEs) / serious adverse events (SAEs) | Up to 2 years.
  Graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE V5.0).

CONTACTS AND LOCATIONS:
Locations (18):
- United States (18):
  - UC San Diego Moores Cancer Center, La Jolla, California
  - University of California, San Francisco (UCSF), San Francisco, California
  - Mount Sinai Comprehensive Cancer Center, Miami Beach, Florida
  - Florida Cancer Specialists, North, St. Petersburg, Florida
  - Florida Cancer Specialists, East, West Palm Beach, Florida
  - Maryland Oncology Hematology, P.A., Brandywine, Maryland
  - Minnesota Oncology Hematology, P.A., Maple Grove, Minnesota
  - Women's Cancer Care Associates, LLC, Albany, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Cincinnati Medical Center, Cincinnati, Ohio
  - Oncology Associates of Oregon, P.C., Eugene, Oregon
  - Northwest Cancer Specialists, P.C., Portland, Oregon
  - Alliance Cancer Specialists, PC, Doylestown, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - Texas Oncology - West Texas, El Paso, Texas
  - Texas Oncology - Gulf Coast, The Woodlands, Texas
  - Virginia Cancer Specialists, P.C., Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Starks DC, Rojas-Espaillat L, Meissner T, Williams CB. Phase I dose escalation study of dual PI3K/mTOR inhibition by Sapanisertib and Serabelisib in combination with paclitaxel in patients with advanced solid tumors. Gynecol Oncol. 2022 Sep;166(3):403-409. doi: 10.1016/j.ygyno.2022.07.005. Epub 2022 Jul 15. PMID 35843739
- See also: Related Info — https://faeththerapeutics.com/